CLINICAL TRIAL: NCT00506623
Title: A Phase Ⅱ Study of Pre-Operative Concurrent Chemoradiotherapy With Capecitabine Plus Irinotecan in Resectable Rectal Cancer.
Brief Title: Preoperative Chemoradiotherapy With Capecitabine Plus Irinotecan in Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS 04-088
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Rectal Neoplasm; Neoadjuvant Therapy
Keywords: Rectal neoplasm; Neoadjuvant therapy; Radiotherapy; Combination chemotherapy; Irinotecan; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — capecitabine-irinotecan combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine, Irinotecan

SUMMARY:
This study is to evaluate the pathologic complete response rate to pre-operative concurrent chemoradiotherapy with capecitabine plus irinotecan in resectable rectal cancer

DETAILED DESCRIPTION:
This study is an open-label, single center, nonrandomized phase II study. Daily fractions of radiotherapy at 1.8 Gy to total of 45 Gy to tumor and draining lymph nodes and followed by a coned-down boost of 5.4 Gy to the tumor were delivered concurrently with chemotherapy.

Chemotherapy starts at day 1 of radiotherapy. Capecitabine is administered orally at a dose of 825 mg/m2 twice daily during weekdays (Monday to Friday) every week during radiotherapy. Irinotecan 40 mg/m2 is given intravenously once a week (D 1, 8, 15, 22 & 29).

Six ± 2 weeks after completion of chemoradiotherapy, curative surgery is performed.

Post-operative chemotherapy with capecitabine will be given to all patients 3-6 weeks after surgery. Capecitabine 1,250 mg/m2 twice daily on days 1-14 every 21 days will be administered for 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum
* Distal margin of tumor located from 0 to 8 cm from anal verge
* Tumor must be clinically resectable by surgery and R0 resection must be most likely
* ECOG performance status 0-2
* No prior chemotherapy, radiotherapy to pelvis, and immunotherapy
* Adequate organ functions
* Patients must sign an informed consent

Exclusion Criteria:

* Malignant disease of the rectum other than adenocarcinoma or arisen from chronic inflammatory bowel disease
* Any unresected synchronous colon cancer
* Any distant metastasis
* Intestinal obstruction or impending obstruction, but decompressing colostomy is permitted
* Any previous or concurrent malignancy other than non-melanoma skin cancer or in situ cancer of uterine cervix
* Any other morbidity or situation with contraindication for chemoradiotherapy
* Patients have history of significant gastric or small bowel resection, or malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may compromise the absorption of capecitabine
* Pregnant or lactating women or patients of childbearing potential not practicing adequate contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-07; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic stage Tumor regression grade | After operation

SECONDARY OUTCOMES:
Toxicity | During chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D., Principal Investigator
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea